CLINICAL TRIAL: NCT04055831
Title: Immune Biomarkers Related to Bone Pathology in Patients With Type 1 Gaucher Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 19-LDRTC-01
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Gaucher Disease Type 1
Keywords: Gaucher disease; Osteoporosis
MeSH Terms: conditions — Gaucher Disease; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, PBMC, and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GD1 subjects with no bone complications: 1. GD1 subjects with no bone complications (n=10)
- GD1 patients with mild bone complication: 2. GD1 subjects with mild bone complications
- GD1 with severe bone complications: 3. GD1 subjects with severe bone complications
- No bone disease: Controls with no known bone disease (n=10)

SUMMARY:
Bone-related problems represent the principal unmet medical need in Gaucher disease (GD). 75% of GD type 1 patients develop skeletal complications, including bone remodeling defects, osteopenia, osteoporosis, marrow infiltration, avascular necrosis, and osteolysis. However, the underlying cellular/molecular basis of bone involvement and related complications in GD are not fully known. Neither are there any bone-specific markers associated with individual bone pathology. Early diagnosis of bone disease is the key issue for planning individual therapy to prevent and reverse bone disease in GD.

DETAILED DESCRIPTION:
This clinical observational study is designed to identify specific biomarkers for bone involvement in patients with GD1 with decreased bone density and/or bone structural abnormalities

Aims:

1. Identify novel immune cell surface and biochemical markers in peripheral blood correlating with bone involvement in GD.
2. Assess the correlation between cytokine levels in peripheral blood and the severity of bone involvement in GD.
3. Assess the relationship between glycosphingolipids accumulation and macrophage activation with specific bone markers and GD severity.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in this study the subject must meet the following criteria

  1. Subject is greater than 16 years old but not older than 90 years
  2. Signed Informed Consent/Assent
  3. Subject is able and willing to sign informed consent or assent
  4. If the subject has GD1, the must have a confirmed diagnosis of Gaucher disease by

     * GCase enzyme activity
     * DNA analysis demonstrating pathogenic variants in the GBA gene

Exclusion Criteria:

* a) Have evidence of hepatitis B, hepatitis C infection or any other chronic infectious disease b) Be pregnant or breastfeeding

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinically confirmed GD1 patients will be stratified based on their disease severity and bone density findings.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Measure biomarkers level in molar/l/h | 18 months
  Bone homeostasis is dependent on the balance of deposition by osteoblasts
  DMP-1, OSCAR, Calcitonin, Lyso-GB1, chitotriosidase, CCL18, osteocalcin, BALP, cathepsin K , TRAP 5, RANKL, OPG, DDK-1, sclerostin, MCP1, IL-2, IL-6, IL-10, SRTH2 and TNF-α
Measure biomarkers level: molar/mg/h | 18 months
  DMP-1, RANK, OSCAR, cathepsin K, OPG

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — Lysosomal and Rare Disorders Research and Treatment Center
Locations (1):
- LDRTC, Fairfax, Virginia, United States

REFERENCES:
- [Derived] Ivanova MM, Dao J, Kasaci N, Friedman A, Noll L, Goker-Alpan O. Wnt signaling pathway inhibitors, sclerostin and DKK-1, correlate with pain and bone pathology in patients with Gaucher disease. Front Endocrinol (Lausanne). 2022 Nov 24;13:1029130. doi: 10.3389/fendo.2022.1029130. eCollection 2022. PMID 36506070